CLINICAL TRIAL: NCT05724017
Title: Determining the Effect of Street Play Intervention on Children's Play Tendencies and Social Problem Solving Levels: I Learn to Solve My Problems by Playing Project
Brief Title: Determining the Effect of Street Play Intervention on Children's Play Tendencies and Social Problem Solving Levels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Atlas University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AtlasU2
Record Dates: First submitted 2023-01-27; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Child Behavior; Child, Only; Playing Role; Play Role; Problem;Learning; Nursing Caries
Keywords: Child; Play; Problem solving; Nursing
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Intervention Model Description: in a single group pretest-posttest research design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Street Games Intervention Group (Experimental): Street Games Intervention Group
  Interventions: Behavioral: Street Games Intervention

INTERVENTIONS:
Behavioral: Street Games Intervention — The children to be included in the study will be grouped in groups of 10 according to their age groups. Groups of 10 people consist of six sessions in total, two days a week for three weeks. Applications will be made in the school garden. In the meetings, games that attract the attention of children will be discussed, suitable games will be played, origami, painting and story sharing will be made. In the study, the independent variable street games intervention will be applied.

SUMMARY:
Determining the Effect of Street Play Intervention on Children's Play Tendencies and Social Problem Solving Levels: I Learn to Solve My Problems by Playing Project

DETAILED DESCRIPTION:
Children are affected from a biopsychosocial point of view, both due to the difficulties and restrictions brought by the pandemic and due to the restriction of their play needs due to their developmental period. It is important to intervene through recreational activities in terms of protecting the health of children. In studies conducted with children, no study has been found that evaluates the effects of street games on playing tendencies and social problem solving levels. This study is unique in that it evaluates the effects of street games on playing tendencies and social problem solving levels and is carried out by undergraduate students. It is important to protect and improve the health of children. As a result of this application planned for children, it is aimed to increase the children's tendency to play and their social problem solving levels with the intervention of street games. It is thought that the stress level of children with an increased tendency to play and problem-solving skills will decrease and the risk of catching diseases will decrease accordingly. In addition, it is predicted that compliance with the treatment and care of physical and mental diseases that develop due to the pandemic process will be easier, and there will be a decrease in the rates of application to treatment institutions and hospitalizations. At least 50 children will also form the sample. Data will be obtained by Personal Information Form (PIF), Playing Tendency Scale, Social Problem Solving Inventory - Short Form (SPSI-SF). The children to be included in the study will be grouped in groups of 10 according to their age groups. Groups of 10 people consist of six sessions in total, two days a week for three weeks. Applications will be made in the school garden. In the last session, children will be asked to fill out a questionnaire consisting of the Playing Tendency Scale, Social Problem Solving Inventory - Short Form (SPSI-SF). In the study, answers will be sought to the question "Is there a difference between children's Playing Tendencies and social problem solving levels before and after the street play intervention application?" The analysis of the data obtained will be done using the SPSS 23.0 (Statictical Package for Social Science) package program. In the evaluation of the data, descriptive statistics such as frequency distribution, mean and standard deviation will be used to define the sample, two-pair test or Wilcoxon peer test will be used according to the parametric test assumptions for the comparison of the group within itself, and the Chi-square test will be used for the analysis of categorical data. 95% significance level (or α=0.05 margin of error) will be used to determine the differences in the analyses. The answers to the open-ended questions will be categorized by the researchers and evaluated as numbers and percentages. As a result of our study, the Effect of Street Games Intervention on Children's Playing Tendencies and Social Problem Solving Levels will be determined and a contribution will be made to the literature. The intervention implemented in this study is expected to guide further studies.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Being a student of the designated school,
* To be enrolled in primary school on the specified dates,
* Ability to read and write,
* Parental consent for the child to participate in the study

Exclusion Criteria:

-Having a barrier to communication,

Removal Criteria:

* Not participating in the intervention for more than 2 weeks,
* The development of a medical condition that interferes with the educational process,
* Transferring to another school,
* The participant's right to withdraw from the research at his/her own request or family

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-02-17 (Estimated); Study Completion 2023-05-17 (Estimated)

PRIMARY OUTCOMES:
Children's Play Tendencies | 4 weeks
  Gaming Trends Scale. The scale is a five-point Likert scale (1= "Not at all like this child, 5= "Completely like this child") and each item is given a score in the range of 1-5. The total score that can be obtained from the scale is between 23 and 115. There are two reverse items (#16 and #22) in the scale.
Social Problem Solving Level | 4 weeks
  Social Problem Solving Inventory - Short Form (SPSI-SF). The lowest score obtained from the scale is 0, and the highest score is 100. High scores indicate a "good level" of social problem solving skills, while low scores indicate a low level of social problem solving skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Atlas University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
I can share it to contribute to other researchers.
Time Frame: 6 months